CLINICAL TRIAL: NCT01257217
Title: A Randomized, Subject-Masked Comparison of Visual Function After Bilateral Implantation of Presbyopia-Correcting IOLs
Brief Title: A Comparison of Visual Function After Bilateral Implantation of Presbyopia-Correcting Intraocular Lenses (IOLs)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M09-051
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-03

CONDITIONS: Cataract
Keywords: Intraocular Lens; Presbyopia; multifocal
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ReSTOR +3 (Experimental): AcrySof® IQ ReSTOR® +3.0 D Multifocal IOL Model SN6AD1 or AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric IOL Model SND1TT, lens assignment and model determined by preoperative keratometric astigmatism, bilateral implantation
  Interventions: Device: AcrySof® IQ ReSTOR® +3.0 D Multifocal IOL Model SN6AD1; Device: AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric IOL Model SND1TT
- Acri.LISA (Active Comparator): Acri.LISA® 366D IOL or Acri.LISA® 466TD Toric IOL, lens assignment determined by preoperative keratometric astigmatism, bilateral implantation
  Interventions: Device: Acri.LISA® 366D IOL; Device: Acri.LISA® 466TD Toric IOL

INTERVENTIONS:
Device: AcrySof® IQ ReSTOR® +3.0 D Multifocal IOL Model SN6AD1 — Multifocal IOL implanted for long-term use over the lifetime of the cataract patient
  Arms: ReSTOR +3
Device: AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric IOL Model SND1TT — Multifocal IOL with extended secondary focal point and astigmatism correction implanted for long-term use over the lifetime of the cataract patient
  Other Names: Models SND1T2, SND1T3, SND1T4, SND1T5, SND1T6
  Arms: ReSTOR +3
Device: Acri.LISA® 366D IOL — Aspheric diffractive IOL with +3.75 D add power implanted for long-term use over the lifetime of the cataract patient
  Arms: Acri.LISA
Device: Acri.LISA® 466TD Toric IOL — Aspheric diffractive IOL with +3.75 D add power and astigmatism correction implanted for long-term use over the lifetime of the cataract patient
  Arms: Acri.LISA

SUMMARY:
The purpose of this study is to evaluate visual and refractive parameters in a series of subjects bilaterally implanted with presbyopia-correcting intraocular lenses (IOLs) during cataract surgery.

DETAILED DESCRIPTION:
Each subject completed a preoperative examination of both eyes, implantation of IOL at the operative visit for each eye, and up to 4 postoperative visits (each eye examined at Day 1-2, with binocular visits at Month 1 and Month 3 after the second implantation). The second implantation occurred within 30 days of the first.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent;
* Able to attend postoperative examinations per protocol schedule;
* Diagnosed with bilateral cataracts;
* Planned cataract removal by phacoemulsification with implantation of an intraocular lens (IOL);
* Preoperative astigmatism ≤ 2.5 diopter;
* Good ocular health, with the exception of cataracts;
* Free of disease(s)/condition(s) listed in the "Caution" section of the AcrySof IQ and Acri.LISA package inserts;
* Able to undergo second eye surgery within one month of the first eye surgery;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Previous corneal surgery;
* Planned multiple procedures during cataract/IOL implantation surgery;
* Any ocular disease and/or condition that may compromise study results;
* Pregnant or planning pregnancy during course of study;
* History of corneal disease (e.g., herpes simplex, herpes zoster keratitis, etc.)
* Diabetic retinopathy;
* Macular degeneration;
* History of retinal detachment;
* Other protocol-defined exclusion criteria may apply.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brand Lead, Surgical, Global Medical Affairs, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from one investigative site located in Spain.
Pre-assignment Details: Of the 31 enrolled participants, 1 exited prior to randomization due to withdrawn consent and 5 discontinued after randomization due to adverse event (1) and protocol deviation (4). This reporting group includes all randomized participants who received IOLs without major deviations and/or surgical complications (efficacy population).
Period: Overall Study
Arm/Group | ReSTOR +3 | Acri.LISA
Started | 15 | 10
Completed | 13 | 10
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized participants who received IOLs without major deviations and/or surgical complications (efficacy population).
Groups:
- Total: Total of all reporting groups
Arm/Group | ReSTOR +3 | Acri.LISA | Total
Number analyzed (Participants) | 15 | 10 | 25
Age, Customized [Number; unit: participants]
  < 21 years | 0 | 0 | 0
  ≥ 21 years | 15 | 10 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 6 | 2 | 8
Region of Enrollment [Number; unit: participants]
  Spain | 15 | 10 | 25

OUTCOME MEASURES:

1. Primary Outcome: Mean Binocular Defocus VA at Month 3
Description: Defocus VA (an indicator of the expected range of vision with a presbyopia-correcting IOL) was tested binocularly with the participant's best spectacle correction using a chart. Lenses of different spherical powers were placed in front of the eyes to produce varying levels of defocus. The VA at each spherical power was measured in logarithm of the minimum angle of resolution (logMAR), with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represents better visual acuity.
Time Frame: Month 3 from second eye implantation
Population: This analysis population includes all subjects who received IOLs without major deviations and/or surgical complications.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR +3 | Acri.LISA
Number analyzed (Participants) | 13 | 10
logMAR
  -5.00 diopter | 0.78 (0.26) | 0.59 (0.18)
  -4.50 diopter | 0.65 (0.18) | 0.45 (0.17)
  -4.00 diopter | 0.58 (0.19) | 0.29 (0.13)
  -3.50 diopter | 0.36 (0.13) | 0.18 (0.14)
  -3.00 diopter | 0.15 (0.07) | 0.11 (0.21)
  -2.50 diopter | 0.04 (0.08) | 0.08 (0.20)
  -2.00 diopter | 0.14 (0.13) | 0.20 (0.18)
  -1.50 diopter | 0.30 (0.11) | 0.33 (0.18)
  -1.00 diopter | 0.23 (0.10) | 0.22 (0.16)
  -0.50 diopter | 0.07 (0.06) | 0.07 (0.11)
  0.00 diopter | -0.02 (0.07) | -0.05 (0.14)
  +0.50 diopter | 0.06 (0.08) | 0.06 (0.18)
  +1.00 diopter | 0.26 (0.11) | 0.21 (0.16)
  +1.50 diopter | 0.54 (0.21) | 0.37 (0.19)
  +2.00 diopter | 0.63 (0.23) | 0.51 (0.16)

2. Secondary Outcome: Best Corrected Visual Acuity (BCVA) Across a Range of Distances at Month 3
Description: Visual acuity (VA) was tested binocularly (both eyes together) with correction in place if needed across a range of distances under well-lit conditions using Early Treatment of Diabetic Retinopathy Study (ETDRS) charts. VA was measured in logarithm of the minimum angle of resolution (logMAR), with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represents better visual acuity.
Time Frame: Month 3 from second eye implantation
Population: This analysis population includes all subjects who received IOLs without major deviations and/or surgical complications.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR +3 | Acri.LISA
Number analyzed (Participants) | 13 | 10
logMAR
  Far distance 4 meters (m) | -0.02 (0.08) | -0.05 (0.15)
  Intermediate 70 centimeters (cm) | 0.39 (0.11) | 0.35 (0.09)
  Intermediate 60 cm | 0.33 (0.10) | 0.35 (0.09)
  Intermediate 50 cm | 0.24 (0.11) | 0.28 (0.11)
  Near 33/40 cm | 0.19 (0.13) | 0.20 (0.15)

3. Secondary Outcome: Uncorrected Visual Acuity Across a Range of Distances at Month 3
Description: VA was tested binocularly unaided across a range of distances under well-lit conditions using Early Treatment of Diabetic Retinopathy Study (ETDRS) charts. VA was measured in logarithm of the minimum angle of resolution (logMAR), with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represents better visual acuity.
Time Frame: Month 3 from second eye implantation
Population: This analysis population includes all subjects who received IOLs without major deviations and/or surgical complications.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR +3 | Acri.LISA
Number analyzed (Participants) | 13 | 10
logMAR
  Far distance 4 meters (m) | 0.14 (0.20) | 0.03 (0.16)
  Intermediate 70 centimeters (cm) | 0.37 (0.15) | 0.27 (0.14)
  Intermediate 60 cm | 0.36 (0.16) | 0.33 (0.12)
  Intermediate 50 cm | 0.29 (0.19) | 0.33 (0.12)
  Near 33/40 cm | 0.27 (0.18) | 0.28 (0.12)

4. Secondary Outcome: Mean Refractive Spherical Equivalent at Month 3
Description: A manifest refraction (vision check) was performed using a 100% contrast ETDRS chart under well-lit conditions. Results were documented for sphere, cylinder and axis readings. The refractive spherical equivalent was calculated according to the formula: sphere + ½ cylinder power. Both eyes contributed to the mean.
Time Frame: Month 3 from second eye implantation
Population: This analysis population includes all subjects who received IOLs without major deviations and/or surgical complications.
Measure: Mean (Standard Deviation); unit: diopter
Arm/Group | ReSTOR +3 | Acri.LISA
Number analyzed (Participants) | 13 | 10
diopter | 0.1 (0.49) | -0.3 (0.49)

5. Secondary Outcome: Mean Radner Reading Speed
Description: Reading performance was measured using the Radner Reading Chart with no correction (without) and with best distance corrective aids (with). Reading speed was measured in words per minute.
Time Frame: Month 3 from second eye implantation
Population: This analysis population includes all subjects who received IOLs without major deviations and/or surgical complications.
Measure: Mean (Standard Deviation); unit: wpm
Groups:
- ReSTOR +3/Without: AcrySof® IQ ReSTOR® +3.0 D Multifocal IOL Model SN6AD1 or AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric IOL, lens assignment and model determined by preoperative keratometric astigmatism, bilateral implantation, without corrective aids
- ReSTOR +3/With: AcrySof® IQ ReSTOR® +3.0 D Multifocal IOL Model SN6AD1 or AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric IOL, lens assignment and model determined by preoperative keratometric astigmatism, bilateral implantation, with corrective aids
- Acri.LISA/Without: Acri.LISA® 366D IOL or Acri.LISA® 466TD Toric IOL, lens assignment determined by preoperative keratometric astigmatism, bilateral implantation, without corrective aids
- Acri.LISA/With: Acri.LISA® 366D IOL or Acri.LISA® 466TD Toric IOL, lens assignment determined by preoperative keratometric astigmatism, bilateral implantation, with corrective aids
Arm/Group | ReSTOR +3/Without | ReSTOR +3/With | Acri.LISA/Without | Acri.LISA/With
Number analyzed (Participants) | 13 | 13 | 10 | 10
wpm | 90.60 (26.82) | 90.46 (22.19) | 109.7 (18.21) | 113.2 (17.80)

6. Secondary Outcome: Patient Reported Outcomes at Month 3
Description: The Visual Task Difficulty Assessment (VISTAS) questionnaire was completed by the subject to assess difficulty in completing everyday tasks that depend on good vision. Tasks were rated using a 1 to 5 point scale, where 1 = no difficulty; 2 = minor difficulty; 3 = moderate difficulty; 4 = major difficulty; 5 = cannot accomplish. Individual scores for each task were averaged to obtain the overall score for each vision type/function. Near vision was defined as less than 50 cm; intermediate vision as 50 cm to 1 m; extended intermediate vision as 90 cm to 4 m; and distant vision as more than 4 m.
Time Frame: Month 3 from second eye implantation
Population: This analysis population includes all subjects who received IOLs without major deviations and/or surgical complications.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ReSTOR +3 | Acri.LISA
Number analyzed (Participants) | 13 | 10
units on a scale
  Near function scale score | 1.78 (0.76) | 1.48 (0.84)
  Intermediate function scale score: number analyzed (Participants) | 2 | 4
  Intermediate function scale score | 1.13 (0.18) | 1.19 (0.38)
  Extended intermediate function scale score: number analyzed (Participants) | 13 | 9
  Extended intermediate function scale score | 1.32 (0.51) | 1.00 (0.00)
  Distant function scale score: number analyzed (Participants) | 6 | 6
  Distant function scale score | 1.08 (0.13) | 1.04 (0.10)

ADVERSE EVENTS:
Description: This analysis group includes all subjects who were randomized (N=17 for ReSTOR+3, N=13 for Acri.LISA) into the study.
Groups:
- ReSTOR +3: AcrySof® IQ ReSTOR® +3.0 D Multifocal IOL Model SN6AD1 or AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric IOL
- Acri.LISA: Acri.LISA® 366D IOL or Acri.LISA® 466TD Toric IOL
Arm/Group | ReSTOR +3 | Acri.LISA
Serious Adverse Events (participants affected / at risk) | 2/17 | 0/13
Other Adverse Events (participants affected / at risk) | 10/17 | 1/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ReSTOR +3 (N=17) | Acri.LISA (N=13)
Macular oedema (Eye disorders) | 1 | 0
Posterior capsule rupture (Eye disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ReSTOR +3 (N=17) | Acri.LISA (N=13)
Conjunctival haemorrhage (Eye disorders) | 2 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Corneal oedema (Eye disorders) | 5 | 1
Corneal oedema/ocular hypertension (Eye disorders) | 1 | 0
Ocular hyperaemia/lacrimation (Eye disorders) | 1 | 0
Retinal cyst (Eye disorders) | 1 | 0
Intraocular pressure abnormal (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.